CLINICAL TRIAL: NCT04171440
Title: Perioperative Outcomes of Robotic Approach for Pancreaticoduodenectomy: a Multi-center, Prospective, Single Arm, Observational Study
Brief Title: Observation of Perioperative Outcomes of Robotic Pancreaticoduodenectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J19102; IRB00219628 (Other: Johns Hopkins Medicine IRB)
Record Dates: First submitted 2019-11-19; First posted 2019-11-21 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Pancreaticoduodenectomy
Keywords: minimally invasive, robotic, surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Minimally Invasive Pancreaticoduodenectomy (Experimental): Patients that undergo pancreaticoduodenectomy through small incisions with state-of-the-art robotic-assisted technology.
  Interventions: Procedure: robotic pancreaticoduodenectomy

INTERVENTIONS:
Procedure: robotic pancreaticoduodenectomy — The robotic pancreaticoduodenectomy is performed through small incisions using robotic-assisted technology. Pancreaticoduodenectomy is the operation that is necessary to remove tumors of the head and neck of the pancreas, lower portion of the bile duct, and the ampulla of Vater.

SUMMARY:
This is a multi-site prospective, single arm, observational study examining the outcomes of robotic pancreaticoduodenectomy.

DETAILED DESCRIPTION:
This is a multi-site prospective, single arm, observational study examining the outcomes of robotic pancreaticoduodenectomy. Adult patients with symptomatic benign, premalignant, or resectable malignant pathologies recommended for resection after multidisciplinary review and have already chosen to have robotic surgery will be evaluated for enrolling into the study.

Relevant operative, postoperative, and pathologic outcomes will be collected prospectively. The well-established enhanced recovery after pancreaticoduodenectomy pathway currently used in our institution will be applied to all patients postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Symptomatic benign, premalignant, or resectable malignant periampullary and pancreatic tumor requiring resection
* Fit to undergo elective pancreaticoduodenectomy after evaluation by the surgical and anesthesiology teams
* Able to consent to participate in the study
* Appropriate for robotic approach as determined by participating surgeons

Exclusion Criteria:

* Arterial (superior mesenteric artery, celiac axis, hepatic artery) or venous involvement (superior mesenteric vein, portal vein) which meets the definition of borderline or unresectable tumor
* Pregnancy
* BMI >40 kg/m2
* Patient requires an additional surgical resection during the index operation (such as hepatectomy or colectomy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | up to 90 days post intervention
  Days from date of intervention to discharge

SECONDARY OUTCOMES:
Time to functional recovery | Day 1 post-intervention to functional recovery
  Days to functional recovery, which requires that all the following are met:
  * Pain controlled on oral analgesics only (Yes/no, only the date when the result first changes from No to Yes will be recorded)
  * Able to maintain ≥50% of required caloric intake
  * No need for intravenous fluids for hydration
  * Return to independent mobility or baseline mobility for those with previous mobility deficits
Number of participants experiencing complications | Day 90 post-intervention
  Number of participants who experience Clavien-Dindo Grade III or higher complications
Operative estimated blood loss | During the surgery
  Blood loss during the surgery (unit: ml)
Number of participants experiencing pancreaticoduodenectomy-specific complications | Day 90 post-intervention
  Number of participants who experience complications including pancreatic fistula, delayed gastric emptying, postoperative bleeding, wound infection, bile leak, chyle leak, other gastrointestinal leakage, re-intervention (radiographic,surgical, endoscopic), 30-day mortality, 90-day mortality.
Pathological outcomes as assessed by Pathological response to neoadjuvant therapy | Day 90-post intervention
  Pathological response to neoadjuvant therapy(if there is any) reported by pathologist reviewing the resected surgical specimen. Pathological outcomes as defined by Protocol for Examination of Specimens from Patients with Carcinoma of the Pancreas (Pancreas Exocrine 4.0.0.1), where: complete response (score 0) is no viable cancer cells; marked response/minimal residual cancer (score 1) is presence of single cells or rare small groups of cancer cells; moderate response (score 2) is residual cancer with evident tumor regression, but more than single cells or rare groups of cancer cells; poor or no response (score 3) is extensive residual cancer with no evident tumor regression.
Survival Outcome | Overall survival is from surgery to last time of follow-up or death, assessed up to 60 months-post intervention.
  Recurrence free outcome is from surgery to recurrence.
Quality of life (QoL) as measured by EQ-5D-3L | EQ-5D-3L will be measured at 2 to 4 weeks and 3 to 6 months-post intervention.
  The EQ-5D-3L questionnaire essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
  The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems.This decision results into a 1-digit number that expresses the level selected for that dimension. Numbers range from 1-3, with a higher number reflected more problems.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'Best imaginable health state' and 'Worst imaginable health state', ranging from 0 to 100. A higher score reflects a worse health state.
Quality of life (QoL) as measured by QLQ-C30 (version 3) | QLQ-C30 will be measured at 2 to 4 weeks and 3 to 6 months-post intervention.
  QLQ-C30 questionnaire includes five functional scales, three symptom scales, a global health status / QoL scale, and six single items. All of the scales and single-item measures range in score from 0 to 100. A higher score represents a higher response level.
Exploratory outcomes | 30 days after the surgery
  Comprehensive complication index (CCI) is calculated using the multiple complication information within 30 days after the surgery. Each complication included in the index will be recorded as yes or no, and a Clavien-Dindo Grade will be recorded for each complication marked as yes.

CONTACTS AND LOCATIONS:
Overall Officials: Jin He, MD,PhD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Atrium Health, Charlotte, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Slankamenac K, Graf R, Barkun J, Puhan MA, Clavien PA. The comprehensive complication index: a novel continuous scale to measure surgical morbidity. Ann Surg. 2013 Jul;258(1):1-7. doi: 10.1097/SLA.0b013e318296c732. PMID 23728278